CLINICAL TRIAL: NCT05339568
Title: A Multicenter, Randomized, Open, Parallel Grouping, Investigator-initiated Study Evaluating the Long-term Benefit of Patients With Locally Advanced/Metastatic Non-small Cell Lung Cancer Followed up Using a Patient-wide Management Platform
Brief Title: Patient's Whole Process Follow-up Management(HOPE-1)
Acronym: HOPE-1
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Jiandong Zhang, Director of Oncology Radiotherapy Department, Qianfoshan Hospital
Other Study IDs: WYKA001
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer; Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platform follow-up cohort: This cohort will be managed and follow-up by patients' whole process follow-up platform. The patients can report the symptoms, get the reminder of the hospital visit, get the reminder of medicine taking, get the information of patients education.
  Interventions: Other: Patients' whole process follow-up and management platform
- Routine follow-up cohort: This cohort will be managed and follow-up by the investigators or nurses. This cohort will take the routine follow-up and management way by the hospital.

INTERVENTIONS:
Other: Patients' whole process follow-up and management platform — Patients' whole process follow-up and management platform is a software for the patients and investigators. This platform will use to collect patients' information when they are out of patients and will provide the patients' education materials.
  Groups: Platform follow-up cohort

SUMMARY:
Our project is going to explore whether management and follow-up of locally advanced/metastatic patients using the patient process management platform can prolong patient survival and improve patient quality of life.

DETAILED DESCRIPTION:
Now, the treatment of NSCLC is diversiform, such as radiation and chemotherapy, targeted therapy, immune therapy, the treatment goal is to reduce symptoms, improve quality of life, prolong life. But as a result of the disease itself has the high risk of metastasis and recurrence. The treatment is often accompanied by a series of complications, if the patients don't get medical assistance in time, it will lead high risk to physical and mental health of patients. In China, the intermittent period of domestic treatment is mainly family recuperation, but due to the lack of medical knowledge or self-management and self-restraint ability of patients, they may forget to take medicine, stop medication without permission due to side effects and other behaviors that do not follow the doctor's advice, the poorly patients' compliance will lead to a significant reduction in the treatment effect. NSCLC are often accompanied by anxiety, fear, insomnia and other symptoms, causing a huge psychological burden on patients and their families, affecting the quality of life. Whole process follow-up in tumor therapy plays an important role , it is the crucial link between medical, nursing, and patients. Patients' whole process follow-up and management is an important part of cancer disease management.

It is helpful to relieve the patients and their families of the bad psychology, reduce the symptoms of patients, improve the patient's compliance behavior, relieve the psychological anxiety of patients, make it actively cooperate with the treatment, reduce complications, improve the quality of life of patients, so as to prolong the life cycle.

Our project is going to explore whether management and follow-up of locally advanced/metastatic patients using the patient process management platform can prolong patient survival and improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the research and voluntarily sign the informed consent form (ICF)
2. Male or female subjects who are over 18 years old (inclusive) at the time of signing the informed consent form.
3. The subject is diagnosed pathologically or cytologically with non-small cell lung cancer(NSCLC).
4. According to the 8th edition of the American Joint Committee on Cancer [AJCC], it is classified as stage IIB, stage III, stage IV NSCLC.
5. Not suitable for radical treatment or refuse surgery.
6. The life expectancy is not less than 3 months.
7. Be able to use a smartphone.

Exclusion Criteria:

1. Patients with mental illness.
2. Presence of any other malignant tumor.
3. Patients who are expected to undergo radical surgery.
4. Currently participating in clinical trials.
5. Subjects who judged by the investigator to be unsuitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll locally advanced/Metastatic NSCLC who are not suitable for radical treatment or refuse surgery.
Sampling Method: Probability Sample
Enrollment: 1268 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2030-04-21 (Estimated); Study Completion 2030-08-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | UP to 96 months
  OS was calculated from the date of randomization to death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 96 months
  PFS was calculated from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 96 months.
Adverse events rate | Up to 96 months
  Adverse events were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0.
Patients' follow-up compliance | Up to 96 months
  Patients' follow-up compliance were assessed by the N of hospital visits according to the doctors' advice every year.
The quality of life | Up to 96 months
  The quality of life were assessed by SF-36，The SF-36 questionnaire consists of 8 section, including physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health, also including reported health transition. The scoring steps: 1 encode the scale 2 credit the scale 3 score conversion(conversion formula=(actual score-the possible lowest score of this section)/the difference between the possible highest score and the possible lowest score of this section).The higher the score conversion, the better the health.
Follow-up satisfaction | Up to 96 months
  Follow-up satisfaction were assessed by the questionnaire. The questionnaire is including 12 questions, where 28 is the worst imaginable satisfaction state and 130 is the best imaginable satisfaction state.

CONTACTS AND LOCATIONS:
Overall Officials: Jiandong ZHANG, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
Not decided to share IPD or not, we will discuss by all the investigators, after discussion, we will update the status.